CLINICAL TRIAL: NCT06827379
Title: Acute Effects of Inspiratory Muscle Training With Different Loads on Peripheral Muscle Metabolism and Autonomic Response in COPD Patients: A Randomized Crossover Trial
Brief Title: Acute Effects of Inspiratory Muscle Training on Peripheral Muscle Metabolism and Autonomic Response in COPD Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Eduardo Eriko Tenório de França, Clinical Professor, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 6.669.065
Record Dates: First submitted 2025-01-30; First posted 2025-02-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Exercise; Performance; Lung diseases.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Lung Diseases

STUDY DESIGN:
Intervention Model Description: This is a crossover, randomized study, blinded to the evaluator and the researcher responsible for the statistical analysis. The study will evaluate the acute effects of IMT on peripheral muscle metabolism and the autonomic response of patients with COPD and its participants will participate in three groups at different times: IMT-S (strength): IMT to gain inspiratory muscle strength; TMI-R (resistance): TMI to improve inspiratory muscle resistance and Sham - Sham of TMI. All participants randomized to the study will participate in the three groups with a minimum interval of 48 hours between participation in each of the groups. Randomization will be performed to find out the sequence of participation in the three groups for all participants. For statistical analysis, intention-to-treat analysis will be employed and groups will be compared using Students t-test, for continuous variables, or chi-square, for categorical variables.
  ANOVA split-plot, repeated measures for prim.
Who Masked: Investigator
Masking Description: Blinding of the evaluator and the researcher responsible for statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IMT-S (strength) (Experimental): Will be individualized according to the MIP achieved in the initial assessment of each patient's inspiratory muscle strength, with the load being equivalent to 60% of the MIP in cmH2O.
  Interventions: Other: IMT-S (strength)
- IMT-R (resistance) (Experimental): Three sets of two minutes of maximum, deep inspirations followed by two minutes of rest between them, totaling six minutes of IMT. The initial load of the equipment for the IMT-R group will also be individualized, equivalent to 30% of the MIP in cmH2O.
  Interventions: Other: IMT-R (resistance)
- Sham (Sham Comparator): Three sets of two minutes of maximum, deep inspirations followed by two minutes of rest between them, totaling six minutes of IMT with a minimum load of 3cmH2O.
  Interventions: Other: Sham - IMT

INTERVENTIONS:
Other: IMT-S (strength) — Composed of 3 sets of 1 minute of maximum, deep inspirations, with 2 minutes of rest between sets, totaling 3 minutes of IMT. The initial load will be individualized according to the MIP, with the load equivalent to 60% of the MIP.
  Arms: IMT-S (strength)
Other: IMT-R (resistance) — Composed of 3 sets of 2 minutes of maximum, deep inspirations, with 2 minutes of rest between sets, totaling 6 minutes of IMT. The load will also be individualized according to the MIP, with the load equivalent to 30% of the MIP.
  Arms: IMT-R (resistance)
Other: Sham - IMT — Composed of 3 sets of 2 minutes of maximum, deep inspirations, with 2 minutes of rest between sets, totaling 6 minutes of IMT with a minimum load of 3cmH2O.
  Arms: Sham

SUMMARY:
The study will evaluate the acute effects of inspiratory muscle training (IMT) on peripheral muscle metabolism and autonomic response in patients with chronic obstructive pulmonary disease (COPD). This is a randomized, crossover study, with blinding of the evaluator and the researcher responsible for the statistical analysis. Participants will be divided into three groups at different times: TMI- strength (F), TMI to gain inspiratory muscle strength; IMT- resistance (R), IMT for improving inspiratory muscle resistance; and TMI sham. All participants randomized in the study will participate in the three groups, with a minimum interval of 48 hours between participation in each group. Randomization will determine the sequence of participation in the three groups for all participants.

For statistical analysis, an intention-to-treat approach will be used, and the groups will be compared using the Student's t test for continuous variables or the chi-square test for categorical variables. A split-plot ANOVA with repeated measures will be used for primary outcomes, and analysis of covariance will be conducted to identify differences between groups using baseline scores as covariates. Effect sizes and confidence intervals will be calculated using eta squared.

It is expected that IMT applied at different loads can promote effects on vascular function, peripheral muscle metabolism and the response of the autonomic nervous system in patients with COPD, which can greatly contribute to the understanding of the physiological effects of this therapy and support its prescription. as a therapeutic intervention in the rehabilitation of patients with pulmonary diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD according to the Global Initiative for COPD (GOLD, 2023);
* Aged 40 years or older and under 75 years;
* Providing both oral and written informed consent.

Exclusion Criteria:

* Inability to perform the IMT protocol and/or functional tests;
* Presence of psychiatric disorders or cognitive impairments, progressive neurological disorders, cancer, or chronic pain;
* Cognitive impairment or inability to understand commands.
* Patients who have experienced any health issue or had a COPD exacerbation in the previous month will also be excluded to ensure that the patient's symptoms are stable.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral vascular function and muscle metabolism | Up to four weeks
  Evaluated using Near Infrared Spectroscopy (NIRS). Tissue perfusion measurement will be performed using an arterial occlusion maneuver. After three minutes of rest to stabilize the initial measurements; [tissue oxygen saturation (StO2) measured in percentage (%), oxyhemoglobin (HbO2) and deoxyhemoglobin (HHb) measured in mmHg], the cuff will be inflated above 250 mmHg up to 280 mmHg , so that the blood flow is completely interrupted, being maintained for a period of five minutes, until the stabilization of the measurements. The variables obtained during the arterial occlusion maneuver will be: StO2 recovery time after occlusion, HHb variation during occlusion and StO2 variation during occlusion. The variables obtained during the exercise will be: variation of HHb and StO2, time to reach the lowest StO2, rate of deoxygenation and reoxygenation and walking economy in relation to HHb and StO2.
Heart rate and R-R interval recordings | Up to four weeks
  Patients will be evaluated in the laboratory at 22 degrees Celsius (°C) with relative humidity between 50-60%. They should avoid stimulants, alcohol and exercise the day before the test and refrain from smoking or using bronchodilators for 6 hours before the test. An electrocardiogram will be recorded via Holter (CARDIOS™, Brazil) using a bipolar DII electrode, with three electrodes placed on the chest after asepsis and trichotomy. Holter software will provide time series data of heart intervals, analyzing heart rate variability (HRV) in both the time and frequency domains. In the time domain, indicators of sympathetic and parasympathetic activity will be calculated. In the frequency domain, the low, high and very low frequency bands will be evaluated, with the ratio between low frequency and high frequency, representing sympathovagal balance.

SECONDARY OUTCOMES:
Subjective perception of effort | Up to four weeks
  The subjective perception of effort will be assessed through the application of the Modified Borg Scale. This is a quantified vertical scale of 0 to 10, where 0 represents no effort and 10 represents maximum effort. Patients will be instructed to choose a single score that reflects their degree of effort at the moment.
Lung function | Up to four weeks
  Spirometry will be performed following the criteria of the American Thoracic Society. All patients will perform at least three maneuvers in a sitting position, using a nose clip and mouthpiece. They will be instructed to perform a maximum inspiration until total lung capacity, followed by a maximum and continuous forced expiration for at least six seconds until reaching the residual volume. The forced expiratory volume in the first second (FEV1) in milliliters (ml), forced vital capacity (FVC) in ml, FEV1/FVC ratio and peak expiratory flow (PEF) in liters per second (L/s) will be determined.
Respiratory muscle function | Up to four weeks
  To assess respiratory muscle function, a PowerBreathe device model (KH2 with Breathelink feedback) will be used. The assessment includes measuring maximum inspiratory pressure (MIP) and respiratory muscle resistance in centimeters of water (cmH2O). Patients will remain seated with a nose clip to prevent air leakage. For the PIM, they will exhale to the residual volume and then perform a maximum inspiration held for at least 1.5 seconds, with up to eight repetitions, with the highest value being recorded. Resistance will be measured in an incremental test, starting with 10 cmH2O for two minutes, adding 10 cmH2O with each cycle. The test will be stopped if the patient fails the task or reports significant discomfort or fatigue. Vital signs such as heart rate, respiratory rate and oxygen saturation will be monitored at all times. Dyspnea and fatigue will be assessed with the Modified Borg Scale before and after each test, with words of encouragement provided to optimize performance.
Thickness and thickening fraction and diaphragmatic mobility | Up to four weeks
  Diaphragmatic ultrasound is a valuable tool for examining the structure and function of the diaphragm, requiring a convex transducer and a linear transducer. The diaphragm is visualized through the window of the apposition zone, appearing as a three-layer structure: a central hypoechoic muscular layer between two hyperechoic membranes. During diaphragm contraction, ultrasound of the apposition zone window shows muscle shortening and thickening, with measurable mobility during quiet breathing. Atrophy and contraction will be assessed by measuring diaphragm thickness and thickening fraction. A high frequency linear transducer will be positioned in the apposition zone and between the 8th and 9th intercostal spaces. Diaphragmatic thickening will be measured at the end of expiration and at the end of inspiration. The thickening fraction will be calculated as: inspiratory thickening minus expiratory thickening times one hundred, divided by the expiratory thickening measured as a percentage.
Echointensity and thickness of the quadriceps femoris | Up to four weeks
  Ultrasonography of the femoral quadriceps will use a linear transducer to capture images transversely over the anterior compartment of the right thigh in B-mode. The patient will be in a semi-Fowler, supine position with knees extended, and muscles relaxed. The transducer will be placed perpendicular to the limb at two-thirds of the distance between the anterior superior iliac spine and lateral knee condyle, marked with a pen. A coupling gel will reduce tissue distortion, and minimal pressure will capture the thickness of the rectus femoris and vastus intermedius. Images will be saved for computer analysis, and the same landmarks will be used in repeated assessments. The echo intensity will be analyzed using a region of interest 50 millimeters (mm) high and wide. A grayscale histogram (0 = black to 255 = white) will determine muscle quality, with higher values indicating potential muscle infiltration or myofibril depletion.
Feeling of dyspnea | Up to four weeks
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used to assess this outcome, measuring the degree of dyspnea during specific daily activities. The mMRC is divided into 4 grades, ranging from 0 (dyspnea with strenuous exercise) to 4 (dyspnea with minimal effort, such as dressing or bathing). This scale is widely used in patients due to its simplicity, ease of use, and correlation with quality of life, prognosis, and distance covered in the six-minute walk test.
Functional capacity | Up to four weeks
  Functional capacity will be assessed using a conventional exercise test and a six-minute walk test. The exercise test, carried out first, involves a progressively increasing effort until exhaustion or limiting symptoms appear. Patients will rest 10 minutes before the test and will receive instructions on running and stopping, as well as the correct use of the modified Borg scale. An ergometric treadmill will be used with a ramp protocol up to the patient's tolerable limit. Throughout the test, a 12-lead electrocardiogram will monitor the patient. Blood pressure, peripheral oxygen saturation and dyspnea and fatigue (modified Borg scale) will be recorded at rest, every 2 minutes and after the test. The test will be completed based on the guidelines of the Brazilian Society of Cardiology, and the total distance covered will be recorded as a measure of functional performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal da Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No